CLINICAL TRIAL: NCT02463565
Title: Assessment of Food Intake in Hospitalized Patients: A Prospective Hospital Survey
Brief Title: Assessment of Food Intake in Hospitalized Patients
Acronym: UN+
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Professor, University Hospital, Geneva
Other Study IDs: Quality control programme
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Undernutrition
Keywords: nutritional assessment; food survey; hospitalized patients; hospital food
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- hospitalized patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Food provision and consumption were assessed for all hospitalized patients over a 24h-period survey. This study is a part of a control quality programme and is performed every 4 years since 1999.

DETAILED DESCRIPTION:
During one day, a team of dieticians assessed food provided, consumed and reasons for non-consumption in all hospitalized patients receiving 3 meals/day. Oral nutritional supplements, supplemental enteral and parenteral nutrition were taken into account. Nutritional needs were calculated according to the ESPEN recommendations.

Amount of energy and proteins provided and consumed were calculated using the nutrient analysis software Winrest (FSI, Noisy-le-grand, France).

In 2012, the presence of healthcare-associated infections was recorded during this study.

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients

Exclusion Criteria:

* Exclusive enteral or parenteral nutrition
* Patients who do not receive three meals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients in all wards
Sampling Method: Non-Probability Sample
Enrollment: 4152 (Actual)
Dates: Start 1998-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hospital food provided, consumed and wasted measured in energy (kcal) and gram of proteins | 24 hours

SECONDARY OUTCOMES:
Percentage of underfed patients | 24 hours
Hospital meal quality assessed by questionnaire | 24 hours
Presence of healthcare-associated infections | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Thibault R, Chikhi M, Clerc A, Darmon P, Chopard P, Genton L, Kossovsky MP, Pichard C. Assessment of food intake in hospitalised patients: a 10-year comparative study of a prospective hospital survey. Clin Nutr. 2011 Jun;30(3):289-96. doi: 10.1016/j.clnu.2010.10.002. Epub 2010 Nov 9. PMID 21067850
- [Background] Dupertuis YM, Kossovsky MP, Kyle UG, Raguso CA, Genton L, Pichard C. Food intake in 1707 hospitalised patients: a prospective comprehensive hospital survey. Clin Nutr. 2003 Apr;22(2):115-23. doi: 10.1054/clnu.2002.0623. PMID 12706127
- [Background] Thibault R, Makhlouf AM, Kossovsky MP, Iavindrasana J, Chikhi M, Meyer R, Pittet D, Zingg W, Pichard C. Healthcare-associated infections are associated with insufficient dietary intake: an observational cross-sectional study. PLoS One. 2015 Apr 29;10(4):e0123695. doi: 10.1371/journal.pone.0123695. eCollection 2015. PMID 25923783
- [Derived] Makhlouf AM, Kossovsky MP, Gurba F, Pautex S, Chikhi M, Pichard C, Genton L. Severity of pain is associated with insufficient energy coverage in hospitalised patients: A cross-sectional study. Clin Nutr. 2019 Apr;38(2):753-758. doi: 10.1016/j.clnu.2018.03.005. Epub 2018 Mar 17. PMID 29588127